CLINICAL TRIAL: NCT01179321
Title: Malnutrition Screening and Intervention in Hospitalised Older Patients: A Randomised Controlled Trial
Brief Title: Malnutrition Screening in Acute Aged Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Wales Hospital, Sydney (Other Government)
Responsible Party: Margaret Holyday, Prince of Wales Hospital
Other Study IDs: malscreen05/185
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2006-03

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Restraint, Physical; Nutrition Therapy

ARMS (2):
- Control (No Intervention)
- Early nutrition intervention (Experimental)
  Interventions: Other: Early referral to Dietitian for assessment and nutrition support

INTERVENTIONS:
Other: Early referral to Dietitian for assessment and nutrition support
  Arms: Early nutrition intervention

SUMMARY:
The purpose of this study is to determine the impact of malnutrition screening and nutrition intervention on acute aged care patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* admitted under a geriatrician into one of 2 acute geriatric medicine wards of the hospital

Exclusion Criteria:

* expected length of stay less than 72 hours
* palliative (not for active treatment)
* unable to be nutritionally assessed (non english speaking, severe dementia/confusion and non cooperative/refused)
* already seen by dietitian during current admission
* enrolled in the study during previous admission

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-04

PRIMARY OUTCOMES:
Length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Margaret M Holyday, B.Sc, Principal Investigator — Prince of Wales Hospital
Locations (1):
- Prince of Wales Hospital, Randwick, New South Wales, Australia